CLINICAL TRIAL: NCT00540930
Title: A Randomized Control Trial of Intravitreal Ranibizumab (Lucentis) for the Prevention of Radiation Maculopathy Following Plaque Radiotherapy for Choroidal Melanoma
Brief Title: Intravitreal Ranibizumab for the Prevention of Radiation Maculopathy Following Plaque Radiotherapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shields, Shields and Associates (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 07-816
Record Dates: First submitted 2007-10-05; First posted 2007-10-08 (Estimated); Last update posted 2007-10-08 (Estimated); Status verified 2007-10

CONDITIONS: Uveal Melanoma; Radiation Retinopathy; Radiation Maculopathy
MeSH Terms: conditions — Uveal Melanoma | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Ranibizumab — Intravitreal Ranibizumab 0.5mg at the time of radioactive plaque insertion
  Other Names: Lucentis

SUMMARY:
Uveal Melanoma is the most common primary intraocular malignancy in adulthood. Eye preserving treatments can deliver equivalent life prognosis in the management of small and medium sized uveal melanomas, as compared to enucleation. Plaque radiotherapy has emerged as the most common eye-preserving treatment in the current management of uveal melanoma, but is complicated by visual loss in approximately 70% of patients at 10 years follow-up. Strategies for the prevention and early treatment of radiation retinopathy/maculopathy need to be developed to improve visual outcomes following plaque treatment. Ranibizumab (Lucentis) is the antigen binding fragment of a recombinant, humanized monoclonal antibody, which inhibits the activity of vascular endothelial growth factor A, a mediator in the development of choroidal neovascularization. Lucentis is commonly used in the eye for eye conditions such as age related macular degeneration. This study will investigate the possible benefit of Anti-VEGF therapy (Lucentis) in reducing the incidence of radiation complications following plaque radiation for uveal melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* new diagnosis of choroidal melanoma
* scheduled for plaque radiotherapy at Wills Eye Health System

Exclusion Criteria:

* Pre-existing retinal disorders (i.e. age-related macular degeneration, diabetic maculopathy, retinal vascular occlusion, macular hole, surface wrinkling retinopathy)
* prior retinal detachment
* media opacities precluding accurate OCT imaging
* history of glaucoma
* pregnancy
* age <18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2007-04; Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of optical coherence (OCT) evidence of macular edema. | 4 months

SECONDARY OUTCOMES:
Grade of macular edema on OCT, visual acuity (LogMAR), and foveal thickness measurement on OCT at follow-up. | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Carol L Shields, MD, Principal Investigator — Wills Eye Institute
Locations (1):
- Wills Eye Institute, Philadelphia, Pennsylvania, United States